CLINICAL TRIAL: NCT02754310
Title: Repeated Versus Varied Simulation Scenarios to Teach Medical Students the Management of a Pediatric Asthma Exacerbation: A Randomized Controlled Study
Brief Title: Repeated Versus Varied Simulation Scenarios to Teach Medical Students the Management of a Pediatric Asthma Exacerbation
Acronym: REVAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilumens (Other)
Responsible Party: Principal Investigator, David Drummond, Dr David Drummond, Ilumens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ILUMENS0001
Record Dates: First submitted 2016-04-26; First posted 2016-04-28 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-03

CONDITIONS: Education, Medical
Keywords: Education, medical; Simulation Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Repeated scenarios (Active Comparator): Participants in the repeated scenario group will learn the management of a pediatric asthma exacerbation on the same scenario repeated three times. The scenario is a pediatric moderate asthma exacerbation not responding to treatment, .
  Interventions: Other: Repeated scenarios
- Varied scenarios (Experimental): Participants in the varied scenarios group will learn the management of a pediatric asthma exacerbation on three different scenarios: a moderate asthma exacerbation, a mild one, and a severe one, for the same length of time than the "repeated scenarios" group. In this group, there is a variation of scenarios.
  Interventions: Other: Variation of scenarios

INTERVENTIONS:
Other: Variation of scenarios — Three different scenarios of pediatric asthma exacerbations: a mild exacerbation, a moderate exacerbation, and a severe exacerbation.
  Arms: Varied scenarios
Other: Repeated scenarios — The same scenario of a moderate pediatric asthma exacerbation is repeated three times.
  Arms: Repeated scenarios

SUMMARY:
Repeated exposure to simulated cases has been shown to improve performance, but repeating the same scenario may impair the ability of learners to transfer their knowledge and skills to slightly different situations. The objective of this study is to compare the use of repeated versus varied simulation cases for teaching the management of pediatric asthma exacerbation to 3rd year medical students.

ELIGIBILITY:
Inclusion Criteria:

* Third year medical students from Paris Descartes and Paris Diderot medical faculties.
* Who are not opposed to participated in the study

Exclusion Criteria:

* Opposition to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-05; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Drummond, MD, Principal Investigator — University Paris René Descartes
Locations (1):
- Département de Simulation iLumens, Université Paris Descartes, Paris, France

REFERENCES:
- [Background] Tofil NM, Peterson DT, Wheeler JT, Youngblood A, Zinkan JL, Lara D, Jakaitis B, Niebauer J, White ML. Repeated versus varied case selection in pediatric resident simulation. J Grad Med Educ. 2014 Jun;6(2):275-9. doi: 10.4300/JGME-D-13-00099.1. PMID 24949131
- [Background] Cook DA, Hamstra SJ, Brydges R, Zendejas B, Szostek JH, Wang AT, Erwin PJ, Hatala R. Comparative effectiveness of instructional design features in simulation-based education: systematic review and meta-analysis. Med Teach. 2013;35(1):e867-98. doi: 10.3109/0142159X.2012.714886. Epub 2012 Sep 3. PMID 22938677
- See also: iLumens is the department of simulation in healthcare of the University Paris Descartes in Paris — http://ilumens.fr

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Varied Scenarios | Repeated Scenarios
Started | 42 | 43
Completed | 42 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varied Scenarios | Repeated Scenarios | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 22 [21 to 22] | 22 [21 to 23] | 22 [21 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Asthma [Count of Participants; unit: Participants] | 2 | 3 | 5
Medical Experience in pediatrics [Count of Participants; unit: Participants] | 3 | 8 | 11
Familiar with low-fidelity manikins [Count of Participants; unit: Participants] | 39 | 40 | 79

OUTCOME MEASURES:

1. Primary Outcome: Management Score on Transfer Scenario n°1
Description: The transfer scenario n°1 is a new scenario that learners face for the first time. It is a pediatric asthma exacerbation rapidly worsening.
  The scale "Asthma exacerbation rapidly worsening" includes different items related to the sequence, the dose, and the administration technique of the treatments. The score ranges between 0 and 10, 10 meaning perfect management of the medical condition. The detailed scale can be found in the supplementary material of the article published here: https://link.springer.com/article/10.1007/s00431-017-3054-1.
Time Frame: One week
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Varied Scenarios | Repeated Scenarios
Number analyzed (Participants) | 42 | 43
units on a scale | 8.3 [7.4 to 10.0] | 8.0 [6.0 to 10.0]

2. Secondary Outcome: Management Score on Transfer Scenario n°2
Description: The transfer scenario n°2 is a new scenario that learners face for the first time. It is a pediatric pneumonia. Students are expected to realize that the child's presentation differs from an asthma exacerbation and should not start short-acting beta agonists nor steroids.
  The scale "Pediatric Pneumonia" includes different items related to the sequence of the treatments administered. The score ranges between 0 and 4, 4 meaning perfect management of the medical condition. The detailed scale can be found in the supplementary material of the article published here: https://link.springer.com/article/10.1007/s00431-017-3054-1.
Time Frame: One week
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Varied Scenarios | Repeated Scenarios
Number analyzed (Participants) | 42 | 43
units on a scale | 3.0 [3.0 to 4.0] | 4.0 [3.0 to 4.0]

3. Secondary Outcome: Management Score on Evaluation Scenario n°1
Description: The evaluation scenario n°1 is a scenario of a moderate asthma exacerbation not responding to treatment, used during the learning phase of both groups (3 times for the group "repetition" and just once for the group "variation").
  The scale "moderate asthma exacerbation" includes different items related to the sequence, the dose, and the administration technique of the treatments. The score ranges between 0 and 16, 16 meaning perfect management of the medical condition. The detailed scale can be found in the supplementary material of the article published here: https://link.springer.com/article/10.1007/s00431-017-3054-1.
Time Frame: One week
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Varied Scenarios | Repeated Scenarios
Number analyzed (Participants) | 42 | 43
units on a scale | 14.1 [13.0 to 16.0] | 15.0 [13.0 to 16.0]

4. Secondary Outcome: Management Score on Evaluation Scenario n°2
Description: The evaluation scenario n°2 is a scenario of a mild asthma exacerbation not responding to treatment, used during the learning phase of the "variation group".The scale "mild asthma exacerbation" includes different items related to the sequence, the dose, and the administration technique of the treatments. The score ranges between 0 and 9, 9 meaning perfect management of the medical condition. The detailed scale can be found in the supplementary material of the article published here: https://link.springer.com/article/10.1007/s00431-017-3054-1.
Time Frame: One week
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Varied Scenarios | Repeated Scenarios
Number analyzed (Participants) | 42 | 43
units on a scale | 9.0 [7.5 to 9.0] | 7.0 [2.0 to 9.0]

5. Secondary Outcome: Management Score on Transfer Scenario n°3
Description: The transfer scenario n°3 is a new scenario that learners face for the first time. It is a severe asthma exacerbation improving before relapsing.The scale "Asthma exacerbation improving then relapsing" includes different items related to the sequence, the dose, and the administration technique of the treatments. The score ranges between 0 and 16, 16 meaning perfect management of the medical condition. The detailed scale can be found in the supplementary material of the article published here: https://link.springer.com/article/10.1007/s00431-017-3054-1.
Time Frame: 4 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Varied Scenarios | Repeated Scenarios
Number analyzed (Participants) | 42 | 43
units on a scale | 13.0 [10.4 to 15.3] | 12.3 [9.8 to 16.0]

6. Secondary Outcome: Management Score on Transfer Scenario n°4
Description: The transfer scenario n°4 is a new scenario that learners face for the first time. It is a pediatric laryngitis. Students are expected to realize that the child's presentation differs from an asthma exacerbation and should not start short-acting beta agonists.
  The scale "Pediatric laryngitis" includes different items related to the sequence and the dose of the treatments provided. The score ranges between 0 and 3, 3 meaning perfect management of the medical condition. The detailed scale can be found in the supplementary material of the article published here: https://link.springer.com/article/10.1007/s00431-017-3054-1.
Time Frame: 4 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Varied Scenarios | Repeated Scenarios
Number analyzed (Participants) | 42 | 43
units on a scale | 2.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0]

7. Secondary Outcome: Management Score on Evaluation Scenario n°1
Description: The evaluation scenario n°1 is a scenario of a moderate asthma exacerbation not responding to treatment, used during the learning phase of both groups (3 times for the group "repetition" and just once for the group "variation") The scale "moderate asthma exacerbation" includes different items related to the sequence, the dose, and the administration technique of the treatments. The score ranges between 0 and 16,16 meaning perfect management of the medical condition. The detailed scale can be found in the supplementary material of the article published here: https://link.springer.com/article/10.1007/s00431-017-3054-1.
Time Frame: 4 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Varied Scenarios | Repeated Scenarios
Number analyzed (Participants) | 42 | 43
units on a scale | 13.6 [11.9 to 15.3] | 13.8 [11.0 to 15.3]

8. Secondary Outcome: Management Score on Evaluation Scenario n°2
Description: The evaluation scenario n°2 is a scenario of a mild asthma exacerbation not responding to treatment, used during the learning phase of the "variation group".
  The scale "mild asthma exacerbation" includes different items related to the sequence, the dose, and the administration technique of the treatments. The score ranges between 0 and 16,16 meaning perfect management of the medical condition. The detailed scale can be found in the supplementary material of the article published here: https://link.springer.com/article/10.1007/s00431-017-3054-1.
Time Frame: 4 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Varied Scenarios | Repeated Scenarios
Number analyzed (Participants) | 42 | 43
units on a scale | 7.5 [6.8 to 9.0] | 7.5 [5.0 to 9.0]

ADVERSE EVENTS:
Arm/Group | Repeated Scenarios | Varied Scenarios
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No